CLINICAL TRIAL: NCT03550287
Title: A Clinical Trial to Evaluate the Effect of a Shiitake Mushroom Extract Supplement on Lipid Profile, Other Cardiovascular Risk Factors and the Microbiota in Subjects With and Moderate Hyperlipidemia
Brief Title: Evaluation of the Effect of a Shiitake Extract on Lipid Profile in Subjects With Moderate Hyperlipidemia
Acronym: Reducol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4813
Record Dates: First submitted 2018-05-08; First posted 2018-06-08 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2018-04

CONDITIONS: Hypercholesterolemia; Hyperlipidemias; Dietary Supplements; Cardiovascular Risk Factor
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental product (Experimental): Dietary supplement (Shiitake extract) in a commercial soup at lunch for 8 weeks.
  Interventions: Dietary Supplement: Experimental product
- Placebo product (Placebo Comparator): Isocaloric placebo (maltodextrin) in a commercial soup at lunch for 8 weeks.
  Interventions: Dietary Supplement: Placebo product

INTERVENTIONS:
Dietary Supplement: Experimental product — 10 g/day
  Arms: Experimental product
Dietary Supplement: Placebo product — 10 g/day
  Arms: Placebo product

SUMMARY:
Effect of a dietary supplement with Shiitake extracts (Lentinula edodes) on lipid profile and other cardiovascular risk factors in subjects with moderate hyperlipidemia without pharmacological treatment.

DETAILED DESCRIPTION:
Prospective, parallel, randomized and double-blind clinical-nutritional study of 8 weeks of duration and 2 study groups (1) Food supplement with extracts of the fungus Shiitake; 2) Placebo supplement with maltodextrin) to evaluate the effect of a food supplement derived from the Shiitake mushroom (Lentinula edodes) on the lipid profile, other cardiovascular risk factors and the intestinal microbiota in subjects with hyperlipidemia moderate without pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 65 years old.
* BMI ≥18.5 and <30 kg/m2.
* Adequate cultural level and understanding for the clinical trial.
* Signed informed consent.
* Cardiovascular risk <10% to 10 years measured by REGICOR.
* Total cholesterol ≥ 200 mg/d and at least 2 factors included in the following list:

  * ≥ 45 years or women ≥ 55 years.
  * Family history of cardiovascular disease (CVD) in first degree male relative less than 55 years of age and less than 65 years in women.
  * HDL cholesterol: men <40 or women <50.
  * Triglycerides ≥ 150mg/dL and <200 mg/dL
  * LDL cholesterol ≥ 130mg/dL and < 160mg/dL
  * Smoker
* Willingness to follow a healthy diet, hyperlipidemic control diet and a diet without stanols, sterols and yeast.
* Social or familiar environment that prevents from accomplishing the dietary treatment

Exclusion Criteria:

* Individuals diagnosed with Diabetes Mellitus type 1.
* Individuals diagnosed with Diabetes Mellitus type 2 on pharmacological treatment (unless it is possible the suspension 30 days before the trials).
* Individuals with dyslipidemia on pharmacological treatment;
* Individuals with hypertension on pharmacological treatment;
* Individuals > 60 years smokers with total cholesterol > 200mg/dL or LDL >130mg/dl.
* Individuals with hypertension on pharmacological treatment uncontrolled.
* Individuals with hyperthyroidism and hypothyroidism on pharmacological treatment uncontrolled.
* Individuals allergic to Shiitake (Lentinula edodes)
* Individuals with chronic diseases (hepatic, kidney, …)
* Individuals receiving at least the preceding 2 months a pharmacological treatment that modifies the lipid profile (for example, statins, fibrates, diuretics, corticosteroids, ADOs);
* Individuals who have participated in the last 6 months in a program or clinical trial to lose weight.
* Smokers wanting to stop to smoke during the period that clinical trial lasts.
* Individuals with mental illness.
* Consume drugs to lose weight during 30 days before starting the study
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Total Cholesterol | Week 0 and 8
  Total Cholesterol

SECONDARY OUTCOMES:
Change from Baseline Lipid Metabolism Parameters | Week 0 and 8
  High Density Lipoprotein
Change from Baseline Lipid Metabolism Parameters | Week 0 and 8
  Low Density Lipoprotein
Change from Baseline Lipid Metabolism Parameters | Week 0 and 8
  Triglycerides
Change from Baseline Lipid Metabolism Parameters | Week 0 and 8
  Apolipoprotein B, Apolipoprotein A1, Pancreatic lipase
Change from Baseline Satiety Hunger Assessment | Week 0 and 8
  Visual Analogue Scale (VAS). 100mm horizontal line anchored at each end with the extremes of the subjective feeling to be quantified. Subjects are instructed to rate the sensation being experienced according to how they define the line.
  e.g., "not at all hungry" (0mm) and "as hungry as I have ever felt" (100mm). Multiple measures are taken at repeated time intervals described below.
Total amount of food consumed in 24h | Week 0 and 8
  24h Food Record Method
Change from Baseline Vitamin D | Week 0 and 8
  Vitamin D
Change from Baseline Anthropometric Parameters | Week 0 and 8
  Weight and Height to calcule BMI in kg/m2
Change from Baseline Anthropometric Parameters | Week 0 and 8
  Waist Circumference
Sensory Perception | Week 4
  Questionnaire of analysis of sensory perception of the food study product. Five questions that are valued on a scale of 0% to 100% asking about the taste and smell of the study product: desire with which the product is taken, taste, smell, consistency and what wait for effectiveness.
Change from Baseline Glucose Parameters | Week 0 and 8
  Glucose
Change from Baseline Inflammation Parameters | Week 0 and 8
  PCR, fibrinogen, IL-6, IL-10, TNFalpha
Adverse Effects | Week 0, 4 and 8
  Gastrointestinal Symptoms (Nausea, Diarrhea, Bloating and other disorders)
Change from Baseline Markers of oxidation | Week 0 and 8
  LDLox

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, PhD, MS, Principal Investigator — Institute for Health Research IdiPAZ
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain